CLINICAL TRIAL: NCT07296367
Title: Examining the Relationship Between Disaster Response Self-efficacy, Psychological Preparedness, and Interdisciplinary Readiness in Physiotherapy Students
Brief Title: Physiotherapy and Disaster
Status: Enrolling by invitation | Type: Observational
Sponsor: Uşak University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor
Other Study IDs: E-60116787-020-789573
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Disaster; Physiotherapist Students
Keywords: Disaster response self-efficacy; Interdisciplinary readiness; Physiotherapy students; Disaster management; Psychological preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physiotherapy students: physiotherapy students studying at different universities

SUMMARY:
The purpose of this observational study is to examine the relationships between disaster response self-efficacy, psychological preparedness for disaster threats, and interdisciplinary readiness levels among undergraduate Physiotherapy and Rehabilitation students. The study will be conducted among students studying in the Physiotherapy and Rehabilitation departments of Pamukkale University, İnönü University, and Alanya Alaaddin Keykubat University in Turkey.

Participants will complete online surveys regarding disaster preparedness while continuing their routine education as part of their active learning. No clinical practice, medical intervention, or experimental procedures will be conducted in the study.

The primary research question of this study is:

Is there a significant relationship between the disaster response self-efficacy, psychological preparedness, and interdisciplinary readiness levels of physiotherapy students? Data will be collected voluntarily via Google Form; students can withdraw from the study at any time. Personal information will not be collected, and all data will be analyzed solely for scientific purposes, in accordance with confidentiality principles. While no medical or physical benefits are expected for participants, the findings are expected to contribute to the development of physiotherapy training curricula for disaster preparedness and crisis management.

The study will commence in December 2025 following ethics committee approval, and the entire process, including data collection, is planned to take approximately six months.

DETAILED DESCRIPTION:
This observational study aims to examine the relationships among physiotherapy students' disaster response self-efficacy, psychological preparedness for disaster threats, and interdisciplinary readiness levels. Data will be collected and analyzed from volunteer participants via an online survey. No experimental interventions, treatments, or clinical procedures will be implemented in the study. Participant safety and data confidentiality will be protected in accordance with ethical principles. The findings are expected to contribute to the development of disaster preparedness regulations in physiotherapy education programs.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student (1st-4th year) in a Physiotherapy and Rehabilitation program at a university in Türkiye
* Being 18 to 25 years of age at the time of participation.
* Reading and providing electronic informed consent on the online form.
* Completing the online questionnaire in full.

Exclusion Criteria:

* Not being enrolled as an undergraduate student in a Physiotherapy and Rehabilitation program, or not being in 1st-4th year.
* Being younger than 18 or older than 25 years.
* Not providing electronic informed consent.
* Completing the survey partially or with clear errors (e.g., missing or invalid responses).
* Duplicate entries detected as the same participant filling in the questionnaire more than once.
* Leaving more than 50% of the items unanswered or providing highly inconsistent response patterns that compromise data reliability.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of undergraduate students studying in Physiotherapy and Rehabilitation departments in Türkiye. Participants will include 1st, 2nd, 3rd, and 4th-year students between the ages of 18 and 25 who voluntarily agree to participate and complete the online informed consent and questionnaire form. Data collection will be carried out through online surveys distributed to students enrolled at Pamukkale University, İnönü University, and Alanya Alaaddin Keykubat University.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Psychological Preparedness Level for Disaster Threats | It will be measured once during data collection.
  * Measurement tool: Psychological Preparedness for Disaster Threats Scale (PPDTS)
  * Variable type: Continuous (Likert total score)
  * Purpose: To determine students' psychological resilience and preparedness levels for disaster situations.

SECONDARY OUTCOMES:
Disaster self-efficacy level | It will be measured once during data collection.
  * Measurement tool: Disaster Response Self-Efficacy Scale (DRESES)
  * Purpose: To assess the perception of competence to respond effectively during a disaster.
Interdisciplinary Readiness Level | It will be measured once during data collection.
  * Measurement tool: Readiness for Interprofessional Learning Scale (RIPLS)
  * Purpose: To determine readiness for collaboration in post-disaster healthcare services.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denzili, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because data is collected entirely on a voluntary basis, protecting participant privacy is a priority. Therefore, there are no plans to share Individual Participant Data (IPD) with third parties.